CLINICAL TRIAL: NCT05622591
Title: Dose Escalation Study to Evaluate the Safety and Tolerability of ELU001 in Pediatric Patients Who Have Relapsed and/or Refractory CBFA2T3::GLIS2 Positive Acute Myeloid Leukemia
Brief Title: ELU001 in Pediatric Subjects Who Have Relapsed and/or Refractory CBFA2T3-GLIS2-positive AML
Acronym: Pediatric AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Funding - no safety issue with Drug; Company Permanently Closed
Sponsor: Elucida Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELU-FRα-AML-1
Record Dates: First submitted 2022-11-08; First posted 2022-11-18 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; AML, Childhood; Relapsed Pediatric AML; Refractory Pediatric AML
Keywords: CBFA2T3-GLIS2; CBFA2T3::GLIS2; Refractory; Folate Receptor alpha; Acute Myeloid Leukemia; ELU001; Exatecan; C'Dot drug conjugate; C-Dot; C'Dot; Childhood; Nanoparticle; Folate Receptor; AML; Relapsed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELU001 (Experimental): Dose Escalation: Escalating doses of ELU001
  Interventions: Drug: ELU001

INTERVENTIONS:
Drug: ELU001 — Folic-acid functionalized C'Dot-Drug-Conjugate (FA-CDC)

SUMMARY:
This research study was planned to focus on a rare type of acute myeloid leukemia (with the subtype CBFA2T3::GLIS2 that overexpresses folate receptor alpha (FRα) (a protein on the surface of leukemia cells)) that has relapsed or is refractory. Relapse means the cancer has come back after treatment. Refractory means the cancer does not respond to treatment.

DETAILED DESCRIPTION:
This study was planned as a Dose Escalation Safety Study to identify the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D). This study will also evaluate the tolerability of ELU001.

ELU001 is not a drug approved by the FDA (Food and Drug Administration) yet.

ELIGIBILITY:
Key Inclusion Criteria:

Patients must meet the following criteria to enroll in this study:

* Infants (>1 month) and children (≤9 years) at time of enrollment.
* Relapsed or refractory CBFA2T3::GLIS2 positive AML
* CNS1 or CNS2 during screening
* Performance Status: Lansky ≥ 50
* Adequate Organ Function including liver, kidney, and heart

Key Exclusion Criteria:

Patients who meet any of the following are not eligible to enroll in this study:

* CNS3 Disease
* AML associated with congenital syndromes such as Down syndrome, Fanconi anemia, Bloom syndrome, Kostmann syndrome or Diamond-Blackfan anemia, or bone marrow failure associated with inherited syndromes.
* Acute promyelocytic leukemia.
* Clinically significant active or chronic corneal disorder, particularly corneal epitheliopathy or any eye disorder that may predispose patient to this condition, or unable to comply with an age-appropriate ophthalmologic examination.
* Prior treatment with folate receptor-targeting anti-cancer agent(s) ≤ 21 days (or 2 half-lives must have elapsed before enrollment, whichever is longer), or received investigational anti-cancer treatment ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, prior to starting study drug, whichever is shorter.

Ages: 1 Month to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of ELU001 | 28 days
  Establish the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of ELU001 in pediatric patients with relapsed or refractory CBFA2T3::GLIS2 positive AML.

SECONDARY OUTCOMES:
Evaluate preliminary anti-leukemic activity of ELU001 | First dose of study drug until 42 days after last cycle.
  Proportion of evaluable patients having achieved at least one of the following
  * Complete Remission per IWG (CRIWG)
  * Complete Remission With Partial Recovery of Platelet Count (CRp)
  * Complete Remission with Incomplete Blood Count Recovery (CRi)
  * Complete Remission for Minimal Residual Disease (CRm)
  Duration of Complete Remission from CRIWG/CR/CRp/CRi to hematological relapse or death from any cause, whichever comes first
Characterize the pharmacokinetics of ELU001 | First dose of study drug until 42 days after last cycle.
  Measure the concentration of ELU001 in the blood.
  This includes - Maximum Observed Concentration (Cmax), Time After Dosing at which Maximum Observed Concentration of Drug is Observed (tmax), Area Under the Curve to the End of the Dosing Period (AUC0-tau), and Area Under the Curve to the Last Measurable Concentration (AUC0-t), will be estimated. Other PK parameters, e.g., Terminal Elimination or Disposition Half-Life (T½), Volume of Distribution (Vd), Clearance Rate (CL), and C'Dot, payload on C'Dot
Characterize the immunogenicity of ELU001 | First dose of study drug until 42 days after last cycle.
  Percent incidence of Anti-Drug Antibodies (ADA) formation in the blood assessed from baseline until End-of-Treatment (EOT).

IPD SHARING:
Plan to Share IPD: No